CLINICAL TRIAL: NCT05844553
Title: Assessment and Validation of a Device for Measuring Hydrogen Peroxide in Exhaled Breath Condensate in Healthy Volunteers
Brief Title: Measuring Hydrogen Peroxide in Exhaled Breath Condensate in HV
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 20IC6380
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Proof Of Concept Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Exhaled breath condensate (EBC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy Volunteers
  Interventions: Device: Measurement of inhaled measuring hydrogen peroxide in exhaled breath

INTERVENTIONS:
Device: Measurement of inhaled measuring hydrogen peroxide in exhaled breath — Participant exhales in to device

SUMMARY:
The purpose of this study is to evaluate the performance of an Exhaled Breath Condensate (EBC) device. EBC measurements can be used for the assessments of lung inflammation in asthma and chronic obstructive pulmonary disease (COPD). Current assessments are based on patient symptoms and simple spirometry tests. Unfortunately, these tests are not directly correlated to lung inflammation in these diseases. Exhaled Breath Condensate (EBC) serves as a simple and non-invasive measurement which can potentially inform clinical decision-making. EBC measures hydrogen peroxide (H2O2) concentrations in exhaled breath and significantly higher concentrations are found in COPD patients. Following a successful pilot study we now want to evaluate the device with real breath samples from healthy volunteers. We want to evaluate the consistency of 3 measurements a month apart.

DETAILED DESCRIPTION:
We aim to recruit 20 healthy volunteers . Our purpose with this study is to evaluate the analytical performance of the device and the data processing and consistency of measurement over 3 measurements a month apart.

Participants will be screened to see if they are suitable for the study. The Screening procedure will take approximately one hour and involve the researcher going through a list of questions related to their health and any medications they are currently taking.

A hard copy of the participant information sheet will be provided at the appointment and participants will be encouraged to ask questions. Participants will then be presented with a consent form..

After the consent form has been signed, the breath collection protocol can then begin.

The handheld breath collection apparatus will be switched on by the researcher and allowed to achieve the correct temperature (1-2 minutes). A sterilised disposable plastic mouthpiece will be fitted. The participant will be asked to hold the breath collection device and breath normally into the plastic mouthpiece for up to 5 minutes .

The researcher will take the instrument and remove the condensed breath sample, place it in a numbered vial and remove it for analysis in the laboratory. Ideally, three samples per participant will be collected, but the participant may withdraw consent at any point.

All samples will be pseudonymised to protect participant confidentiality. The individual results of the analysis will be made available to the participants. If requested. Three successive measurements will be made at monthly intervals in each individual healthy volunteer requiring them to visit the Hospital on three occasions.

ELIGIBILITY:
Inclusion Criteria:

non-smokers Healthy individuals, free of significant disease.

* Given written informed consent prior to participation in the study including all of its procedures.
* Comply with the requirements and restrictions listed in the consent form.
* Male or female subject aged 18-65 years at screening.
* Able to complete the study and all measurements.
* Able to read, comprehend, and write at a sufficient level to complete study related materials

Exclusion Criteria:

Subjects will not be eligible if any of the following apply: -

* A history of recreational drug use or allergy which in the opinion of the investigators contra-indicates their participation.
* Participation within 3 months in any other study testing a new molecular entity or drug or involving invasive procedures.
* Those, in the opinion of the investigator, who may prove non-compliant with study procedures.
* History of an upper or lower respiratory infection (including coryza) within 3 weeks of baseline assessments (assessments and entry could be deferred.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial Clinical Respiratory Research Unit (ICRRU), St Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Exhaled Breath Measurement: Patient Exhales into the device
  Measurement of inhaled measuring hydrogen peroxide in exhaled breath: Participant exhales from device
Period: Overall Study
Arm/Group | Exhaled Breath Measurement
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Healthy subjects
Groups:
- Exhaled Breath Measurement: Patient inhales from device
  Measurement of inhaled measuring hydrogen peroxide in exhaled breath: Participant exhales from device
Arm/Group | Exhaled Breath Measurement
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20

OUTCOME MEASURES:

1. Primary Outcome: Hydrogen Peroxide in Exhaled Breath Condensate
Description: Volunteer holds the device and breathes through the mouthpiece normally for a maximum of 5 minutes.
Time Frame: 6 months circa
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Exhaled Breath Measurement
Number analyzed (Participants) | 20
µM | 0.101 (0.110)

ADVERSE EVENTS:
Time Frame: 6 months circa
Arm/Group | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT05844553/Prot_000.pdf